CLINICAL TRIAL: NCT01977976
Title: A Randomized Controlled Trial on the Effect of Endometrial Injury on Improving Ongoing Pregnancy Rate in Subfertile Women Undergoing in Vitro Fertilization Treatment
Brief Title: RCT on the Effect of Endometrial Injury on Ongoing Pregnancy Rate in Subfertile Women Undergoing IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yeung Wing Yee Tracy, Associate Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TY03
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Subfertility
Keywords: Endometrial injury; Pipelle; Implantation; Ongoing pregnancy rate; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial Aspirate (EA) group (Experimental): Endometrial aspirate by pipelle
  Interventions: Procedure: Endometrial aspiration by pipelle
- Control group (No Intervention): No intervention prior to scheduled IVF

INTERVENTIONS:
Procedure: Endometrial aspiration by pipelle — Endometrial aspiration by pipelle is to be performed on LH+7 in the cycle preceding scheduled IVF treatment
  Arms: Endometrial Aspirate (EA) group

SUMMARY:
Implantation failure remains one of the major factors limiting success in IVF treatment. It was postulated that the local injury to endometrium induces secretions of cytokines and growth factors such as leukemia inhibitory factor, interleukin-11, and heparin-binding EGF-like growth factor which enhance decidualisation and facilitate implantation. It may also up-regulate the gene expressions related to endometrial receptivity and optimize the endometrial development. In stimulated cycles, local injury to the proliferative endometrium has been postulated to delay endometrial development thereby inducing synchronicity between endometrium and embryo stage and facilitate implantation (Zhou et al, 2008; Almog et al, 2010; Gnainsky et al, 2010) The aim of the study is to determine whether endometrial injury by endometrial biopsy in mid-secretory phase of the preceding cycle would improve the on-going pregnancy rate in subfertile women undergoing IVF treatment.

DETAILED DESCRIPTION:
Consecutive women attending subfertility clinic at Queen Mary Hospital, University of Hong Kong who are scheduled for IVF treatment will be recruited. Women who have normal uterine cavity will be randomized into study and control groups in 1 to 1 ratio according to a computer-generated randomization list. Patients will be stratified according to the first or repeated cycle.

For patients in the study group, in the cycle immediately preceding the scheduled IVF treatment, LH surge will be determined by daily serum LH level starting from 18 days before the next expected period. LH surge is defined as an elevation of LH to 2 times the level of the average of the previous 3 days and the absolute level of the LH should be more than or equal to 20 IU/L. Women randomized into the study group will have endometrial biopsy performed by pipelle 7 days after the LH surge (LH+7) and they will be instructed to use non-hormonal means of contraception during that cycle. All patients will then proceed to IVF treatment in the next cycle as scheduled. They will receive standard ovarian stimulation according to the departmental protocol and have a maximum of two embryos replaced 2 days after the oocyte retrieval. On-going pregnancy rates between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing IVF for tubal, unexplained or male factor subfertility
* Normal uterine cavity as shown on saline sonogram / hysteroscopy done at baseline

Exclusion Criteria:

* Presence of hydrosalpinx
* Presence of endometrial polyp or fibroid distorting uterine cavity
* IVF cycles carried out for preimplantation genetic diagnosis
* Use of donor gametes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10-12 weeks gestation
  Ongoing pregnancy rate per fresh embryo transfer

SECONDARY OUTCOMES:
implantation rate | 4 weeks after embryo transfer
  number of gestation sac on pelvic scan per number of embryo transferred

OTHER OUTCOMES:
Clinical pregnancy rate | 4 weeks after embryo transfer
  Presence of at least one fetal heart pulsation per fresh embryo transfer 4 weeks after transfer

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Yeung, MRCOG, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yeung TW, Chai J, Li RH, Lee VC, Ho PC, Ng EH. The effect of endometrial injury on ongoing pregnancy rate in unselected subfertile women undergoing in vitro fertilization: a randomized controlled trial. Hum Reprod. 2014 Nov;29(11):2474-81. doi: 10.1093/humrep/deu213. Epub 2014 Sep 8. PMID 25205759